

Statistical Analysis Plan (TFL shells):

| | SPONSOR: |
|----------|----------------------------------------|
| | CicloMed |
| ſ | PROTOCOL NUMBER: |
| | CPX-POM-001 |
| STA | TISTICAL ANALYSIS PLAN<br>(TFL shells) |
| Author: | |
| Version: | Version 2.0 |
| Date: | 03Nov2021 |



**Statistical Analysis Plan (TFL shells):** 

Version 2.0 / 03Nov2021

## **Cover and signature pages**

| Sponsor: | CicloMed |
|---|---|
| Protocol Number: | CPX-POM-001 |
| Study Title: | A Phase 1, First-in-Human, Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients with Advanced Solid Tumors |
| Document Version No | Version 2.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorize its approval.

| Name and Date are no | Name and Date are not required if electronic signatures are used. Do not resize boxes. | | |
|---|---|---|---|
| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
| | Principal<br>Biostatistician II | | |



Statistical Analysis Plan (TFL shells):

| Name and Date are not required if electronic signatures are used. Do not resize boxes. | | | |
|---|---|---|---|
| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
| | Medical Advisor | | |

| lame and Date are | me and Date are not required if electronic signatures are used. Do not resize boxes. | | |
|---|---|---|---|
| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
| | Chief Scientific<br>Officer<br>CicloMed LLC | | |



Statistical Analysis Plan (TFL shells):


## **Table of Contents**

| Cover and signature pages | 2 |
|---|---|
| Table of Contents | 4 |
| Tables 14.1 | 9 |
| Table 14.1-1.1 - Patients disposition (All Patients Enrolled) - Dose Escalation | 9 |
| Table 14.1-1.2 - Patients disposition (All Patients Enrolled) – Expansion | 11 |
| Table 14.1-2.1 - Number (%) of Patients in the Analysis Populations (All Patients Enrolled) - Dose Escalation | 14 |
| Table 14.1-2.2 - Number (%) of Patients in the Analysis Populations (All Patients Enrolled) - Expansion | 15 |
| Table 14.1-3.1 - Summary of Demographic and Baseline Characteristics (Safety Population) - Dose Escalation | 16 |
| Table 14.1-3.2 - Summary of Demographic and Baseline Characteristics (Safety Population) - Expansion | 20 |
| Table 14.1-4.1 - Important Protocol Deviations (Safety Population) - Dose Escalation | 21 |
| Table 14.1-4.2 - Important Protocol Deviations (Safety Population) - Expansion | 21 |
| Table 14.1-5.1.1 - Disease Characteristics (Safety Population) - Dose Escalation | 22 |
| Table 14.1-5.1.2 - Disease Characteristics (Safety Population) - Expansion | 26 |
| Table 14.1-5.2.1 - Other Medical History (Safety Population) - Dose Escalation | 27 |
| Table 14.1-5.2.2 - Other Medical History (Safety Population) - Expansion | 28 |
| Table 14.1-5.3.1 - Concomitant Diseases (Safety Population) - Dose Escalation | 28 |
| Table 14.1-5.3.2 - Concomitant Diseases (Safety Population) - Expansion | 28 |
| Table 14.1-6.1.1 - Prior Medications by Therapeutic Class and Preferred Term (Safety Population) - Dose Escalation | 29 |
| Table 14.1-6.1.2 - Prior Medications by Therapeutic Class and Preferred Term (Safety Population) - Expansion | 30 |
| Table 14.1-6.2.1 - Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population) - Dose Escalation | |
| Table 14.1-6.2.2 - Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population) - Expansion | 30 |
| Table 14.1-7.1 - Overall Exposure to Study Drug and Drug Compliance (Safety Population) - Dose Escalation | 31 |
| Table 14.1-7.2 - Overall Exposure to Study Drug and Drug Compliance (Safety Population) - Expansion | 32 |
| Tables 14.2 | 33 |
| Table 14.2-1.1 - Patients who have had at least one other post-baseline tumor assessment (Efficacy Population) Dose Escalation | |
| Table 14.2-2.1 - Summary of Patients Responses (Efficacy Population) - Dose Escalation | 34 |
| Table 14.2-3.2 - Recurrence-Free Survival (RFS) (Efficacy Population) - Expansion | 36 |
| Table 14.2-4.2 - Overall Survival (OS) (Efficacy Population) - Expansion | 37 |
| Table 14.2-5.2 - Patients who Undergo Radical Cystectomy (Efficacy Population) - Expansion | 38 |
| Tables 14.3 | 39 |
| Table 14.3-1.0 - Dose-Limiting Toxicity (DLT) (Safety Population) - Dose Escalation | 39 |
| Table 14.3-1.1.1 - Overview of Adverse Events (Safety Population) - Dose Escalation | 40 |



Statistical Analysis Plan (TFL shells):

| Table 14.3-1.1.2 - Overview of Adverse Events (Safety Population) - Expansion41 |
|---|
| Table 14.3-1.2.1 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Dose Escalation42 |
| Table 14.3-1.2.2 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Expansion |
| Table 14.3-1.3.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Dose Escalation |
| Table 14.3-1.3.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Expansion |
| Table 14.3-1.4.1 - Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Dose Escalation |
| Table 14.3-1.4.2 - Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Expansion |
| Table 14.3-1.5.1 - Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Dose Escalation44 |
| Table 14.3-1.5.2 - Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Expansion45 |
| Table 14.3-1.6.1 - Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population) - Dose Escalation |
| Table 14.3-1.6.2 - Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population) - Expansion45 |
| Table 14.3-1.7.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population) - Dose Escalation |
| Table 14.3-1.7.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population) - Expansion46 |
| Table 14.3-1.8.1 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity (Safety Population) - Dose Escalation |
| Table 14.3-1.8.2 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity (Safety Population) - Expansion48 |
| Table 14.3-1.9.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population) - Dose Escalation |
| Table 14.3-1.9.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population) - Expansion |
| Table 14.3-2.1.1.1 - Summary of Hematology Laboratory Data (Safety Population) - Dose Escalation |
| Table 14.3-2.1.1.2 - Summary of Hematology Laboratory Data (Safety Population) - Expansion50 |
| Table 14.3-2.1.2.1 - Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population) - Dose Escalation |
| Table 14.3-2.1.2.2 - Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population) - Expansion |
| Table 14.3-2.1.3.1 - On-treatment Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Dose Escalation |
| Table 14.3-2.1.3.2 - On-treatment Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Expansion |



Statistical Analysis Plan (TFL shells):

| Table 14.3-2.1.4.1 - Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population) - Dos<br>Escalation | |
|---|---|
| Table 14.3-2.1.4.2 - Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population) - Expansion | 56 |
| Table 14.3-2.2.1.1 - Summary of Clinical Chemistry Laboratory Data (Safety Population) - Dose Escalation | 57 |
| Table 14.3-2.2.1.2 - Summary of Clinical Chemistry Laboratory Data (Safety Population) - Expansion | 57 |
| Table 14.3-2.2.2.1 - Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population) - Dose Escalation | 57 |
| Table 14.3-2.2.2.2 - Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety<br>Population) - Expansion | 58 |
| Table 14.3-2.2.3.1 - On-treatment Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety<br>Population) - Dose Escalation | |
| Table 14.3-2.2.3.2 - On-treatment Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety<br>Population) - Expansion | |
| Table 14.3-2.2.4.1 - Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population) - Dose Escalation | 59 |
| Table 14.3-2.2.4.2 - Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population) - Expansion | 59 |
| Table 14.3-2.3.1.1 - Summary of Coagulation Laboratory Data (Safety Population) - Dose Escalation | 60 |
| Table 14.3-2.3.1.2 - Summary of Coagulation Laboratory Data (Safety Population) - Expansion | 60 |
| Table 14.3-2.3.2.1 - Outside of Normal Range - Shift Table for Coagulation Laboratory Parameters (Safety Population) - Dose Escalation | 60 |
| Table 14.3-2.3.2.2 - Outside of Normal Range - Shift Table for Coagulation Laboratory Parameters (Safety Population) - Expansion | 61 |
| Table 14.3-2.4.1.1 - Summary of Thyroid Panel Laboratory Data(Safety Population) - Dose Escalation | 62 |
| Table 14.3-2.4.1.2 - Summary of Thyroid Panel Laboratory Data(Safety Population) - Expansion | 62 |
| Table 14.3-2.4.2.1 - Outside of Normal Range - Shift Table for Thyroid Panel Laboratory Parameters (Safety Population) - Dose Escalation | 62 |
| Table 14.3-2.4.2.2 - Outside of Normal Range - Shift Table for Thyroid Panel Laboratory Parameters (Safety Population) - Expansion | 63 |
| Table 14.3-2.5.1 - Summary of Other Laboratory Data (Safety Population) - Dose Escalation | 64 |
| Table 14.3-2.5.2 - Summary of Other Laboratory Data (Safety Population) - Expansion | 65 |
| Table 14.3-3.1.1 - Summary of Vital Signs (Safety Population) - Dose Escalation | 66 |
| Table 14.3-3.1.2 - Summary of Vital Signs (Safety Population) - Expansion | 66 |
| Table 14.3-3.2.1 - Summary of Abnormal Vital Signs (Safety Population) - Dose Escalation | 67 |
| Table 14.3-3.2.2 - Summary of Abnormal Vital Signs (Safety Population) - Expansion | 70 |
| Table 14.3-4.1.1 - Summary of ECG Parameters (Safety Population) - Dose Escalation | 71 |
| Table 14.3-4.1.2 - Summary of ECG Parameters (Safety Population) - Expansion | 71 |
| Table 14.3-4.2.1 - Summary of Abnormal ECG Intervals (Safety Population) - Dose Escalation | 72 |
| Table 14.3-4.2.2 - Summary of Abnormal ECG Intervals (Safety Population) - Expansion | 74 |
| Table 14.3-4.3.1 - Shift Table for ECG Overall Interpretation (Safety Population) - Dose Escalation | 75 |



### Statistical Analysis Plan (TFL shells):

| Table 14.3-4.3.1 - Shift Table for ECG Overall Interpretation (Safety Population) - Expansion | 76 |
|---|---|
| Figures | 77 |
| Figure 14.2-4.2 - Recurrence-Free Survival (RFS) (Efficacy Population) – Expansion | 77 |
| Figure 14.2-5.2 - Overall Survival (OS) (Efficacy Population) - Expansion | 78 |
| Listings | 79 |
| Listing 16.2.1-1.1.1 - Preface to Inclusion and Exclusion Criteria - Dose Escalation | 79 |
| Listing 16.2.1-1.1.2 - Preface to Inclusion and Exclusion Criteria - Expansion | 80 |
| Listing 16.2.1-1.2.1 - List of Failed Inclusion and Exclusion Criteria (All Patients) - Dose Escalation | 81 |
| Listing 16.2.1-1.2.2 - List of Failed Inclusion and Exclusion Criteria (All Patients) - Expansion | 81 |
| Listing 16.2.1-2.1 - Patient Disposition (Safety Population) - Dose Escalation | 82 |
| Listing 16.2.1-2.2 - Patient Disposition (Safety Population) - Expansion | 83 |
| Listing 16.2.2.1 - Protocol Deviations (Safety Population) - Dose Escalation | 84 |
| Listing 16.2.2.2 - Protocol Deviations (Safety Population) - Expansion | 84 |
| Listing 16.2.3.1 - Analysis Populations (Safety Population) - Dose Escalation | 85 |
| Listing 16.2.3.2 - Analysis Populations (Safety Population) - Expansion | 85 |
| Listing 16.2.4-1.1 - Demographic and Baseline Characteristics (Safety Population) - Dose Escalation | 86 |
| Listing 16.2.4-1.2 - Demographic and Baseline Characteristics (Safety Population) - Expansion | 87 |
| Listing 16.2.4-2.1 - Pregnancy Test Results (Safety Population) - Dose Escalation | 88 |
| Listing 16.2.4-2.2 - Pregnancy Test Results (Safety Population) - Expansion | 88 |
| Listing 16.2.4-3.1 - Cancer History (Safety Population) - Dose Escalation | 89 |
| Listing 16.2.4-4.1 - Prior Cancer Therapies (Safety Population) - Dose Escalation | 90 |
| Listing 16.2.4-5.1 - Medical History and Concomitant Disease (Safety Population) - Dose Escalation | 91 |
| Listing 16.2.4-5.2 - Medical History and Concomitant Disease (Safety Population) - Expansion | 92 |
| Listing 16.2.4-6.1 - Cardiac Function (Safety Population) - Dose Escalation | 93 |
| Listing 16.2.4-6.2 - Cardiac Function (Safety Population) - Expansion | 93 |
| Listing 16.2.4-7.1 - Ophthalmologic Exam (Safety Population) - Dose Escalation | 94 |
| Listing 16.2.4-8.1.1 - Prior and Concomitant Medications (Safety Population) - Dose Escalation | 95 |
| Listing 16.2.4-8.1.2 - Prior and Concomitant Medications (Safety Population) - Expansion | 96 |
| Listing 16.2.4-8.2.2 - Chemotherapy (Safety Population) - Expansion | 97 |
| Listing 16.2.4-9.1 - Surgeries and Procedures (Safety Population) - Dose Escalation | 98 |
| Listing 16.2.4-9.2 - Surgeries and Procedures (Safety Population) - Expansion | 99 |
| Listing 16.2.5-1.1 - Treatment Administration (Safety Population) - Dose Escalation | 100 |
| Listing 16.2.5-1.2 - Treatment Administration (Safety Population) - Expansion | 101 |
| Listing 16.2.5-2.1 - Infusion Interruption (Safety Population)- Dose Escalation | 102 |
| Listing 16.2.5-2.2 - Infusion Interruption (All Patients Enrolled) - Expansion | 102 |
| Listing 16.2.5-3.1 - Drug Exposure (Safety Population) - Dose Escalation | 103 |
| Listing 16.2.5-3.2 - Drug Exposure (Safety Population) - Expansion | 103 |



Statistical Analysis Plan (TFL shells):

| Listing 16.2.6-1.1 - RECIST Target Lesions (Efficacy Population) - Dose Escalation | 104 |
|---|---|
| Listing 16.2.6-2.1 - RECIST Non-Target Lesions (Efficacy Population) - Dose Escalation | 105 |
| Listing 16.2.6-3.1 - RECIST response (Efficacy Population) - Dose Escalation | 106 |
| Listing 16.2.6-4.1 - Tumor Marker (Efficacy Population) - Dose Escalation | 107 |
| Listing 16.2.6-5.2 - Evaluable TURBT Results (Efficacy Population) - Expansion | 108 |
| Listing 16.2.6-6.2 - Radical Cystectomy (Efficacy Population) - Expansion | 109 |
| Listing 16.2.6-7.2 - Determination of Recurrence and Survival (Efficacy Population) - Expansion | 110 |
| Listing 16.2.6-8.2 - Recurrence-Free Survival and Overall Survival (Efficacy Population) - Expansion | 111 |
| Listing 16.2.7-1.1 - Dose-Limiting Toxicity (Safety Population) - Dose Escalation | 112 |
| Listing 16.2.7-2.1 - Adverse Events (Safety Population) - Dose Escalation | 113 |
| Listing 16.2.7-2.2 - Adverse Events (Safety Population) - Expansion | 113 |
| Listing 16.2.7-3.1 - Serious Adverse Events (Safety Population) - Dose Escalation | 113 |
| Listing 16.2.7-3.2 - Serious Adverse Events (Safety Population) - Expansion | 114 |
| Listing 16.2.7-4.1 - Adverse Events Leading to Discontinuation (Safety Population) - Dose Escalation | 114 |
| Listing 16.2.7-4.2 - Adverse Events Leading to Discontinuation (Safety Population) - Expansion | 114 |
| Listing 16.2.7-5.1 - Adverse Events Leading to Death (Safety Population) - Dose Escalation | 115 |
| Listing 16.2.7-5.2 - Adverse Events Leading to Death (Safety Population) - Expansion | 115 |
| Listing 16.2.8-1.1 - Patients Laboratory Profile: Hematology (Safety Population) - Dose Escalation | 116 |
| Listing 16.2.8-1.2 - Patients Laboratory Profile: Hematology (Safety Population) - Expansion | 117 |
| Listing 16.2.8-2.1 - Patients Laboratory Profile: Clinical Chemistry (Safety Population) - Dose Escalation | 117 |
| Listing 16.2.8-2.2 - Patients Laboratory Profile: Clinical Chemistry (Safety Population) - Expansion | 117 |
| Listing 16.2.8-3.1 - Patients Laboratory Profile: Coagulation (Safety Population) - Dose Escalation | 118 |
| Listing 16.2.8-3.2 - Patients Laboratory Profile: Coagulation (Safety Population) - Expansion | 118 |
| Listing 16.2.8-4.1 - Patients Laboratory Profile: Thyroid Panel (Safety Population) - Dose Escalation | 118 |
| Listing 16.2.8-4.2 - Patients Laboratory Profile: Thyroid Panel (Safety Population) - Expansion | 119 |
| Listing 16.2.8-5.1 - Patients Laboratory Profile: Urinalysis (Safety Population) - Dose Escalation | 120 |
| Listing 16.2.8-5.2 - Patients Laboratory Profile: Urinalysis (Safety Population) - Expansion | 120 |
| Listing 16.2.9-1.1 - Vital Signs (Safety Population) - Dose Escalation | 121 |
| Listing 16.2.9-1.2 - Vital Signs (Safety Population) - Expansion | 122 |
| Listing 16.2.9-2.1 - ECG Results (Safety Population) - Dose Escalation | 123 |
| Listing 16.2.9-2.2 - ECG Results (Safety Population) - Expansion | 124 |
| Listing 16.2.9-3.1 - Digital Holter Monitoring (Safety Population) - Dose Escalation | 125 |



**Statistical Analysis Plan (TFL shells):** 


### **Tables 14.1**

Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Table 14.1-1.1 - Patients disposition (All Patients Enrolled) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM [D2] mg/m^2 N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM [D6] mg/m^2 N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Cycle 1 [n (%)] | | | | | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [a] [c] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 [n (%)] | | | | | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [b] [c] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

#### <repeat until last cycle>

Percentages are based on the number of patients enrolled.

- [a] A patient completed Cycle 1 if s/he attended visit Day 10 (if Cycle 1 was not the last cycle).
- [b] A patient completed Cycle 2 (or any next cycle) if s/he attended visit Day 6 (if Cycle 2 or any next cycle was not the last cycle).
- [c] A patient completed the Last Cycle if s/he attended the last visit of the cycle (visit Day 10 for Cycle 1 or visit Day 6 for Cycle 2 or any next cycle) and if s/he attended the final visit at least 22 days after the first dose in the last cycle.
- [d] Calculated as [(Date of end of study Date of first dose) + 1]/30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-1.1 - Patients disposition (All Patients Enrolled) - Dose Escalation

| | CPX-POM | CPX-POM | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM<br>[D4] mg/m^2 | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2 |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2<br>N=X | | | | | |
| | N=X | | | N=X | | | N=X |
| Reason for end of study [n (%)] | | | | | | | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dose Limitimg Toxicity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy | | | | | | | |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Attended the follow-up visit (Day 28) [n (%)] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Time on study (Months) [d] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

Percentages are based on the number of patients enrolled.

- [a] A patient completed Cycle 1 if s/he attended visit Day 10 (if Cycle 1 was not the last cycle).
- [b] A patient completed Cycle 2 (or any next cycle) if s/he attended visit Day 6 (if Cycle 2 or any next cycle was not the last cycle).
- [c] A patient completed the Last Cycle if s/he attended the last visit of the cycle (visit Day 10 for Cycle 1 or visit Day 6 for Cycle 2 or any next cycle) and if s/he attended the final visit at least 22 days after the first dose in the last cycle.

[d] Calculated as [(Date of end of study - Date of first dose) + 1]/30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Table 14.1-1.2 - Patients disposition (All Patients Enrolled) - Expansion

| | Cisplatin<br>ineligible<br>N=X | Chemotherapy<br>eligible<br>N=X | Overall<br>N=X |
|---|---|---|---|
| Cycle 1 [n (%)]) | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [a] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 [n (%)]) | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 3 [n (%)] [d] | | XX (XX.X) | XX (XX.X) |
| Treated | | XX (XX.X) | XX (XX.X) |
| Completed the cycle [c] | | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of patients enrolled.

- [a] A patient completed Cycle 1 if s/he attended visit Day 6.
- [b] A patient completed Cycle 2 if s/he attended visit Day 26.
- [c] A patient completed Cycle 3 if s/he attended visit Day 48.
- [d] Applicable to Chemotherapy eligible group only.
- [e] A patient completed the study if s/he completed 2 cycles (cisplatin-ineligible patients) or 3 cycles (chemotherapy eligible patients) and had radical cystectomy.
- [f] Calculated as [(Date of end of study Date of first dose) + 1]/30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-1.2 - Patients disposition (All Patients Enrolled) - Expansion

| | Cisplatin<br>ineligible<br>N=X | Chemotherapy<br>eligible<br>N=X | Overall<br>N=X |
|---|---|---|---|
| ompleted end of treatment visit (Day 42 or Day 64) n (%)] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| iscontinued from treatment [n (%)] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| eason for discontinuation from the treatment [n %)] | | | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dose Limitimg Toxicity | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ndergone radical cystectomy (Day 56 or Day 78) [n %)] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ompleted the study [e] | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ompleted at least one follow-up visit [n (%)] | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of patients enrolled.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>a] A patient completed Cycle 1 if s/he attended visit Day 6.

<sup>[</sup>b] A patient completed Cycle 2 if s/he attended visit Day 26.

<sup>[</sup>c] A patient completed Cycle 3 if s/he attended visit Day 48.

<sup>[</sup>d] Applicable to Chemotherapy eligible group only.

<sup>[</sup>e] A patient completed the study if s/he completed 2 cycles (cisplatin-ineligible patients) or 3 cycles (chemotherapy eligible patients) and had radical cystectomy.

<sup>[</sup>f] Calculated as [(Date of end of study - Date of first dose) + 1]/30.4375.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.1-1.2 - Patients disposition (All Patients Enrolled) - Expansion

| | Cisplatin<br>ineligible<br>N=X | Chemotherapy<br>eligible<br>N=X | Overall<br>N=X |
|---|---|---|---|
| Reason for end of study [n (%)] | | | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Time on study (Months) [f] | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX |
| Median | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX |

Percentages are based on the number of patients enrolled.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>a] A patient completed Cycle 1 if s/he attended visit Day 6.

<sup>[</sup>b] A patient completed Cycle 2 if s/he attended visit Day 26.

<sup>[</sup>c] A patient completed Cycle 3 if s/he attended visit Day 48.

<sup>[</sup>d] Applicable to Chemotherapy eligible group only.

<sup>[</sup>e] A patient completed the study if s/he completed 2 cycles (cisplatin-ineligible patients) or 3 cycles (chemotherapy eligible patients) and had radical cystectomy.

<sup>[</sup>f] Calculated as [(Date of end of study - Date of first dose) + 1]/30.4375.



Statistical Analysis Plan (TFL shells):


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-2.1 - Number (%) of Patients in the Analysis Populations (All Patients Enrolled) - Dose Escalation

| | CPX-POM 30<br>mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM<br>[D5] mg/m^2<br>N=X<br>n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Safety Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Efficacy Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of enrolled patients.

The Safety population includes all patients who have received at least one dose of CPX-POM.

The Efficacy population includes all patients who have received at least one dose of CPX-POM, had RECIST measurable disease at baseline and had at least one other post-baseline tumor assessment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- For the safety population, patients are displayed based on the actually received treatment.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-2.2 - Number (%) of Patients in the Analysis Populations (All Patients Enrolled) - Expansion

| | Cisplatin<br>ineligible<br>N=X<br>n (%) | Chemotherapy eligible N=X n (%) | Overall<br>N=X<br>n (%) |
|---|---|---|---|
| Safety Population | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Efficacy Population | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of enrolled patients.

The Safety population includes all patients who have received at least one dose of CPX-POM.

The Efficacy population includes all patients who have received at least one dose of CPX-POM and had available tumor tissue at baseline and at the time of radical cystectomy.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• For the safety population, patients are displayed based on the actually received treatment.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-3.1 - Summary of Demographic and Baseline Characteristics (Safety Population) - Dose Escalation

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2<br>N=X | [D2] mg/m^2<br>N=X | [D3] mg/m^2<br>N=X | [D4] mg/m^2<br>N=X | [D5] mg/m^2<br>N=X | [D6] mg/m^2<br>N=X | [D7] mg/m^2<br>N=X |
| Acc [a] (rearc) | | | | | | | |
| Age [a] (years) | XX | XX | XX | XX | XX | XX | XX |
| n<br>Mana | | | | | | | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Age group [n (%)] | | | | | | | |
| < 65 years | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ≥ 65 years | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Sex [n (%)] | | | | | | | |
| Male | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Female | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Race [n (%)] | | | | | | | |
| White | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Asian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| American Indian or Alaska Native | XX (XX.X) | XX (XX.X) | XX (XX . X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other Pacific Islander | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other Pacific Islander Other | , | , , | , , | , , | , , | XX (XX.X) | XX (XX.X) |
| Orliet | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | $\wedge \wedge (\wedge \wedge \cdot \wedge)$ | ΛΛ (ΛΛ•Λ) |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] Body mass index (BMI)  $(kg/m^2) = Weight (kg) / (Height (m))^2$ .

<sup>[</sup>c] The denominator is the number of females in each dose group.

<sup>[</sup>d] Body Surface Area (BSA)  $(m^2) = 0.007184 \times Weight (kg)^0.425 \times (Height (m))^0.725 (Dubois formula).$ 



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-3.1 - Summary of Demographic and Baseline Characteristics (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| <pre>Female of child beari potential [n (%)] [c]</pre> | | | | | | | |
| Able to bear childr | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Premenarche | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Post Menopausal | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Sterile - of child bearing age | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Country [n (%)] | | | | | | | |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Height (cm) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] Body mass index (BMI)  $(kg/m^2)$  = Weight (kg) / (Height (m))\*\*2.

<sup>[</sup>c] The denominator is the number of females in each dose group.

<sup>[</sup>d] Body Surface Area (BSA)  $(m^2) = 0.007184 \times Weight (kg)^0.425 \times (Height (m))^0.725 (Dubois formula)$ .



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-3.1 - Summary of Demographic and Baseline Characteristics (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM [D2] mg/m^2 N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Weight (kg) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| BMI [b] (kg/m^2) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| BSA [d] (m^2) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] Body Mass Index (BMI)  $(kg/m^2) = Weight (kg) / (Height (m))^2$ .

<sup>[</sup>c] The denominator is the number of females in each dose group.

<sup>[</sup>d] Body Surface Area (BSA)  $(m^2) = 0.007184 \times Weight (kg)^0.425 \times (Height (m))^0.725 (Dubois formula)$ .



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


### Table 14.1-3.1 - Summary of Demographic and Baseline Characteristics

| | ( | Safety Populat | ion) - Dose Es | scalation | | | |
|---|---|---|---|---|---|---|---|
| | CPX-POM<br>30 mg/m^2 | CPX-POM<br>[D2] mg/m^2 | CPX-POM<br>[D3] mg/m^2 | CPX-POM<br>[D4] mg/m^2 | CPX-POM<br>[D5] mg/m^2 | CPX-POM<br>[D6] mg/m^2 | CPX-POM<br>[D7] mg/m^2 |
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| ECOG [n (%)] | | | | | | | |
| 0 (Fully active) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <pre>1 (Unable to perform physically<br/>strenuous activity but ambulatory<br/>and able to carry out work of a</pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| light or sedentary nature) 2 (Ambulatory and capable of all selfcare but unable to carry out any work activities) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 (Capable of only limited selfcare) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 (Completely disabled) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

- [a] Age at Screening.
- [b] Body Mass Index (BMI)  $(kg/m^2) = Weight (kg) / (Height (m))^2$ .
- [c] The denominator is the number of females in each dose group.
- [d] Body Surface Area (BSA)  $(m^2) = 0.007184 \times Weight (kg)^0.425 \times (Height (m))^0.725 (Dubois formula).$

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

### Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.1-3.2 - Summary of Demographic and Baseline Characteristics (Safety Population) - Expansion

Replicate of Table 14.1-3.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.1-4.1 - Important Protocol Deviations (Safety Population) - Dose Escalation

| Protocol Deviations Category | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D2] mg/m^2<br>N=X<br>n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Any Important Protocol Deviations | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <pre>Inclusion / Exclusion Criteria INCL01 <cont.></cont.></pre> | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| Prohibited Medications | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <cont.></cont.> | | | | | | | |

A patient could be counted under more than one category.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Categories are from the protocol deviations criteria form, the table only shows examples.
- A last column with the header 'CPX-POM All Doses' will also be displayed.

Table 14.1-4.2 - Important Protocol Deviations (Safety Population) - Expansion

#### Replicate of Table 14.1-4.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Table 14.1-5.1.1 - Disease Characteristics (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2 | CPX-POM [D2] mg/m^2 | CPX-POM [D3] mg/m^2 | CPX-POM [D4] mg/m^2 | CPX-POM [D5] mg/m^2 | CPX-POM [D6] mg/m^2 | CPX-POM [D7] mg/m^2 |
|---|---|---|---|---|---|---|---|
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| Primary Tumor Site [n (%)] | | | | | | | |
| Bladder Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Breast Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Colon Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Gastric Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Head and Neck Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Liver | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Ovarian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Prostate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Time Since First Diagnosis of | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Disease Stage at Screening Vis | sit Date? [n (%)] | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Presence of Metastases? [n (% | ) ] | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Table 14.1-5.1.1 - Disease Characteristics (Safety Population) - Dose Escalation

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| Extent of Current Metastatic disease | Э | | | | | | |
| Abdomen/Viscera? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adrenals? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Bladder? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Bone? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Bone Marrow? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Chest Wall? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| CNS/Brain? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Kidnet? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Table 14.1-5.1.1 - Disease Characteristics (Safety Population) - Dose Escalation

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| Lungs? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Liver? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lymp Nodes? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pancreas? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Peritoneal? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Plura? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stomach? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Spleen? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


### PROGRAMMING NOTES:

A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

# Table 14.1-5.1.2 - Disease Characteristics (Safety Population) - Expansion

| | Cisplatin ineligible N=X n (%) | Chemotherapy<br>eligible<br>N=X<br>n (%) | Overall<br>N=X<br>n (%) |
|---|---|---|---|
| | 11 (0) | 11 (0) | 11 (0) |
| Dose expansion Arm | | | |
| Cisplatin-ineligible patient | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Chemotherapy-eligible patient | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason [a] | | | |
| Creatinine clearance < 60 mL/min | XX (XX.X) | | XX (XX.X) |
| <pre>Heart failure (NYHA class &gt;=III)</pre> | XX (XX.X) | | XX (XX.X) |
| Grade >=2 hearing loss | XX (XX.X) | | XX (XX.X) |
| Grade >=2 neuropathy | XX (XX.X) | | XX (XX.X) |
| Other | XX (XX.X) | | XX (XX.X) |
| Screening eGFR (mL/min/1.73m2) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX |
| Median | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX |

eGFR = estimated Glomerular Filtration Rate.

[a] Applicable to Cisplatin ineligible group only .

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.1-5.2.1 - Other Medical History (Safety Population) - Dose Escalation

| System Organ Class/<br>Preferred Term | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM<br>[D5] mg/m^2<br>N=X<br>n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| At least one other previous condition? | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| System Organ Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- The Primary System Organ Classes are presented by alphabetical order and the Preferred Terms are sorted within Primary System Organ Classes by alphabetical order.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.1-5.2.2 - Other Medical History (Safety Population) - Expansion

Replicate of Table 14.1-5.2.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.1-5.3.1 - Concomitant Diseases (Safety Population) - Dose Escalation

Replicate of Table 14.1-5.2.1

#### PROGRAMMING NOTES:

• Add footnote: `Events with both start and end dates missing were considered as concomitant.'

Replicate of Table 14.1-5.3.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Table 14.1-6.1.1 - Prior Medications by Therapeutic Class and Preferred Term (Safety Population) - Dose Escalation

| Therapeutic Class/<br>Preferred Term | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| At least one prior medication? | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Therapeutic Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Therapeutic Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

A prior medication is a medication whose end date is before the date of first CPX-POM dose.

If there was more than one prior medication reported under the same Therapeutic Class and Preferred Term, the patient was counted only once under that Therapeutic Class and Preferred Term. If there was more than one prior medication reported under the same Therapeutic Class, the patient was counted only once under that Therapeutic Class.

WHO-DRUG version Version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- The Therapeutic Classes are presented by alphabetical order and the Preferred Terms are sorted within Therapeutic Classes by alphabetical order.
- A medication / therapy can appear within more than one Therapeutic Class.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



Statistical Analysis Plan (TFL shells):


Table 14.1-6.1.2 - Prior Medications by Therapeutic Class and Preferred Term (Safety Population) - Expansion

#### Replicate of Table 14.1-6.1.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.1-6.2.1 - Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population) - Dose Escalation

#### Replicate of Table 14.1-6.1.1

#### PROGRAMMING NOTES:

- Update foootnote: replace 'A prior medication is a medication whose end date is before the date of first CPX-POM dose' by 'A concomitant medication is a medication that started before the date of first dose and stopped on (or is ongoing after) the date of first dose OR a medication whose start date is either the same as (or after) the date of first dose'.
- Update 'At least one prior medication' by 'At least one concomitant medication'.
- The Therapeutic Classes are presented by alphabetical order and the Preferred Terms are sorted within Therapeutic Classes by alphabetical order.
- A medication / therapy can appear within more than one Therapeutic Class.

Table 14.1-6.2.2 - Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population) - Expansion

#### Replicate of Table 14.1-6.2.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.1-7.1 - Overall Exposure to Study Drug and Drug Compliance (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-PO<br>[D7]<br>mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Study Drug Exposure (days) [a] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| tudy Drug Exposure (mg) [b] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] The CPX-POM exposure expressed in days is calculated from the dose administration entered in the database as (last dose taken date - first dose taken date + 1) + 16.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] The CPX-POM exposure expressed in mg is calculated from the dose per m^2 entered in the database as the sum of all (dose per m^2 x Body Surface Area), using Body Surface Area calculated at baseline for Cycle 1 and Cycle 2 dose administrations, and calculated on Day 1 of every other treatment cycle from Cycle 3 dose administration.



**Statistical Analysis Plan (TFL shells):** 


#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.

Table 14.1-7.2 - Overall Exposure to Study Drug and Drug Compliance (Safety Population) - Expansion

Replicate of Table 14.1-7.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


### **Tables 14.2**

Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.2-1.1 - Patients who have had at least one other post-baseline tumor assessment (Efficacy Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| At least one other post-baseline tumor assessment | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary Tumor Type [n (%)] | | | | | | | |
| Bladder Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Breast Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Carcinomatosis | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Colon Cancer | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| COION Cancer | | | | | | XX (XX.X) | XX (XX.X) |

\e\c/

Note: A subject with overall response but no detailed tumor assessments is considered as having tumor assessment in this table.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.2-2.1 - Summary of Patients Responses (Efficacy Population) - Dose Escalation

| Visit/<br>Type of Response | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Cycle 2-Day 1 Visit | | | | | | | |
| Target Lesion Response [n (%)] | | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Target Lesion Response [n (% | | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Overall Response [n (%)] | | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page 34 of 125

### <repeat for Day 1 visit of each cycle from Cycle 3 to last Cycle number over all patients>

Percentage was based on the number of patients with non-missing tumor assessment at each visit.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.2-3.2 - Recurrence-Free Survival (RFS) (Efficacy Population) - Expansion

| | Cisplatin<br>ineligible<br>N=X | Chemotherapy<br>eligible<br>N=X | Overall<br>N=X |
|---|---|---|---|
| Included in the analysis | XX | XX | XX |
| No. of events (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No. of censored observations (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Recurrence-Free Survival Time (Months) [a] | | | |
| Minimum | XX.X | XX.X | XX.X |
| 25% quartile | XX.X | XX.X | XX.X |
| Median (95% CI) [b] | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| 75% quartile | XX.X | XX.X | XX.X |
| Maximum | XX.X | XX.X | XX.X |
| KM probability estimate for Recurrence-Free Survival rate (95% CI) [c] | | | |
| 3 months | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| 6 months | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| 12 months | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |

<sup>[</sup>a] Kaplan-Meier estimates.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- If the median time to event has not been reached, present as "NR (xx.x, xx.x)" [replacing xx.x with '-' if there is no upper or lower confidence limit].
- Time categories to be updated dependent upon the data.

<sup>[</sup>b] 95% confidence interval (CI) for median recurrence-free survival is calculated using the Brookmeyer and Crowley method.

<sup>[</sup>c] Probability estimates are based upon Kaplan-Meier estimates and 95% CI use the log-log transformation.


**Statistical Analysis Plan (TFL shells):** 


Table 14.2-4.2 - Overall Survival (OS) (Efficacy Population) - Expansion

Replicate of Table 14.2-3.2

## PROGRAMMING NOTES:

• Replace 'Recurrence-Free Survival' by 'Overall Survival' in the table and footnotes.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.2-5.2 - Patients who Undergo Radical Cystectomy (Efficacy Population) - Expansion

| | Cisplatin<br>ineligible<br>N=X<br>n (%) | Chemotherapy<br>eligible<br>N=X<br>n (%) | Overall N=X n (%) |
|---|---|---|---|
| Number of patients who undergo radical cystectomy | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



**Statistical Analysis Plan (TFL shells):** 


## **Tables 14.3**

Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-1.0 - Dose-Limiting Toxicity (DLT)
 (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM<br>[D3] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D4] mg/m^2<br>N=X<br>n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Number of patients with at least one DLT | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

MedDRA version <version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-1.1.1 - Overview of Adverse Events (Safety Population) - Dose Escalation

| | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Number of patie with | | | | | | | |
| at least one: | | | | | | | |
| AE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| TEAE * | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| TEAE leading to discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE leading to | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| discontinuation | | | | | | | |
| Serious TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Serious related TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>\*</sup> A treatment-emergent adverse events (TEAE) is defined as an adverse event that started on or after the first dose of CPX-POM administration.

MedDRA version version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

- "Leading to discontinuation" is derived from action taken = permanently discontinued.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-1.1.2 - Overview of Adverse Events
(Safety Population) - Expansion

Replicate of Table 14.3-1.1.1

- Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.
- Replace footnote '\* A treatment-emergent adverse events (TEAE) is defined as an adverse event that started on or after the first dose of CPX-POM administration' by '\* A treatment-emergent adverse events (TEAE) is defined as an adverse event that started on or after the first dose of CPX-POM administration and before the date of the last CPX-POM dose + 30 days or the date of start of a new anti-cancer therapy or the date of radical cystectomy, whichever occurs first.'



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001 --- DELIVERY TYPE --- Page 1 of X
Extract date: DDMMMYYYY

Table 14.3-1.2.1 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Dose Escalation

| System Organ Class | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM [D2] mg/m^2 N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM [D7] mg/m^2 N=X |
|---|---|---|---|---|---|---|---|
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Number of patients with at least one TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

If there was more than one TEAE reported under the same System Organ Class and Preferred Term, the patient was counted only once under that System Organ Class and that Preferred Term. If there was more than one TEAE reported under the same System Organ Class, the patient was counted only once under that System Organ Class.

MedDRA version <version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

- The System Organ Classes are presented by decreasing frequency (within the total column all CPX-POM doses groups combined) and the Preferred Terms within a System Organ Class are presented by decreasing frequency (within the total column all CPX-POM doses groups combined).
- A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-1.2.2 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) - Expansion

## Replicate of Table 14.3-1.2.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.3-1.3.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred

Term

(Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.2.1

#### PROGRAMMING NOTES:

• Adjust footnote to mention 'related TEAE' instead of 'TEAE'.

Table 14.3-1.3.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

(Safety Population) - Expansion

## Replicate of Table 14.3-1.3.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-1.4.1 - Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

(Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.2.1

#### PROGRAMMING NOTES:

• Adjust footnote to mention 'serious TEAE' instead of 'TEAE'.

Table 14.3-1.4.2 - Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred

Term

(Safety Population) - Expansion

## Replicate of Table 14.3-1.4.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.3-1.5.1 - Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and
Preferred Term
(Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.2.1

## PROGRAMMING NOTES:

• Adjust footnote to mention 'serious related TEAE' instead of 'TEAE'.



Statistical Analysis Plan (TFL shells):


Table 14.3-1.5.2 - Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and
Preferred Term
(Safety Population) - Expansion

## Replicate of Table 14.3-1.5.1

#### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.3-1.6.1 - Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ

Class and Preferred Term

(Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.2.1

#### PROGRAMMING NOTES:

- "Leading to discontinuation" is derived from Did AE lead to study discontinuation? = Yes.
- Adjust footnote to mention 'TEAE leading to discontinuation' instead of 'TEAE'.

Table 14.3-1.6.2 - Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ
Class and Preferred Term
(Safety Population) - Expansion

## Replicate of Table 14.3-1.6.1

#### PROGRAMMING NOTES:



Statistical Analysis Plan (TFL shells):


Table 14.3-1.7.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events Leading to Discontinuation by System
Organ Class and Preferred Term
(Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.2.1

## PROGRAMMING NOTES:

- "Leading to discontinuation" is derived from Did AE lead to study discontinuation? = Yes.
- Adjust footnote to mention 'related TEAE leading to discontinuation' instead of 'TEAE'.

Table 14.3-1.7.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events Leading to Discontinuation by System
Organ Class and Preferred Term
(Safety Population) - Expansion

## Replicate of Table 14.3-1.7.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY


Filename: (Specify file name.rtf)

Table 14.3-1.8.1 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity

(Safety Population) - Dose Escalation

--- DELIVERY TYPE ----

Dose group: CPX-POM 30 mg/m $^2$  (N=X) System Organ Class Any CTC Preferred Term CTC grade 1 CTC grade 2 CTC grade 3 CTC grade 4 CTC grade 5 grade Maximal severity n (%) n (%) n (%) n (%) n (%) n (%) Number of patients with any TEAE XX (XX.X) XX (XX.X)XX (XX.X)XX (XX.X) XX (XX.X) XX (XX.X)System Organ Class #1 Preferred Term #1 XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X)XX (XX.X)Preferred Term #2 XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X)Preferred Term #3 XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X)<et.c> XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)System Organ Class #2 Preferred Term #1 XX (XX.X) XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)Preferred Term #2 XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Preferred Term #3 XX (XX.X) XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X)XX (XX.X) <etc> XX (XX.X)XX (XX.X)XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X)

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

- Display all severities even if there are no patients.
- The System Organ Classes are presented by alphabetically.
- 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-1.8.2 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity (Safety Population) - Expansion

### Replicate of Table 14.3-1.8.1

#### PROGRAMMING NOTES:

• Include three groups: 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.

Table 14.3-1.9.1 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population) - Dose Escalation

## Replicate of Table 14.3-1.8

#### PROGRAMMING NOTES:

• Adjust footnote to mention 'related TEAE' instead of 'TEAE'.

Table 14.3-1.9.2 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population) - Expansion

## Replicate of Table 14.3-1.9.1

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-2.1.1.1 - Summary of Hematology Laboratory Data (Safety Population) - Dose Escalation

Laboratory Parameter: Hemoglobin (unit)

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| BAS [a] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| C1 TRT D4 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Change from BAS | | | | | | | |
| to C1 TRT D4 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<repeat for Cycle 1 Day 10 visit>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 4 visit> <for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit>

[a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)



**Statistical Analysis Plan (TFL shells):** 


#### PROGRAMMING NOTES:

• Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count and Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils).

• A last column with the header 'CPX-POM All Doses' will also be displayed.

Table 14.3-2.1.1.2 - Summary of Hematology Laboratory Data (Safety Population) - Expansion

Replicate of Table 14.3-2.1.1.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-2.1.2.1 - Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population) - Dose Escalation

Dose group: CPX-POM 30 mg/m^2 (N=X)

| | | | I | Baseline [a] va | lue | |
|---|---|---|---|---|---|---|
| Parameter/ | Value | Low | Normal | High | Low/High* | |
| Visit | at Visit | n (%) | n (%) | n (%) | n (%) | Total |
| Hemoglobin (unit) | | | | | | |
| C1 TRT D4 (N**=XX) | Low | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | High | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Low/High* | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| C1 TRT D10 (N**=XX) | Low | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | High | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Low/High* | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 4 visit>
<for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit>
<repeat for all doses groups>

Percentage was based on the number of patients present at each visit with non-missing results for the considered parameter.

- \* Includes patients with Low or High results. \*\* Denominator of the percentage.
- [a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

- Repeat for all doses groups, including 'CPX-POM All Doses'.
- Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count and Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils).



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.1.2.2 - Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.2.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Table 14.3-2.1.3.1 - On-treatment Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Dose Escalation

| Parameter/<br>Worst NCI-CTCAE grade | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM<br>[D3] mg/m^2<br>N=X<br>n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Hemoglobin (unit) | | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hematocrit (unit) | | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

## <repeat for the other hematology parameters>

A patient with multiple results for a parameter will only be counted once under the maximum NCI-CTCAE grade for this parameter. Laboratory ranges are based on NCI-CTCAE version 4.03.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

- Repeat for all gradable hematology parameters.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.1.3.2 - On-treatment Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Expansion

Replicate of Table 14.3-2.1.3.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Table 14.3-2.1.4.1 - Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population) - Dose Escalation

Dose group:  $CPX-POM 30 mg/m^2 (N=X)$ 

| | | | | | Worst NCI-C | TCAE grade | | |
|---|---|---|---|---|---|---|---|---|
| | Baseline | Normal | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Missing | Total |
| Parameter | grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hematocrit (unit) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 4 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Missing | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Hemoglobin (unit) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 4 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Missing | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

## <repeat for the other hematology parameters>

A patient with multiple results for a parameter will only be counted under the maximum NCI-CTCAE grade for this parameter. Laboratory ranges are based on NCI-CTCAE version 4.03.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

- Repeat for all doses groups, including 'CPX-POM All Doses'.
- Repeat for all gradable hematology parameters.



Statistical Analysis Plan (TFL shells):


Table 14.3-2.1.4.2 - Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.4.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.2.1.1 - Summary of Clinical Chemistry Laboratory Data (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.1.1

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase, Corrected Calcium

Table 14.3-2.2.1.2 - Summary of Clinical Chemistry Laboratory Data (Safety Population) - Expansion

Replicate of Table 14.3-2.1.1.2

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase, Corrected Calcium

Table 14.3-2.2.2.1 - Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population) - Dose Escalation

#### Replicate of Table 14.3-2.1.2.1

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase, Corrected Calcium



Statistical Analysis Plan (TFL shells):


Table 14.3-2.2.2.2 - Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population) - Expansion

## Replicate of Table 14.3-2.1.2.2

## PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase, Corrected Calcium

Table 14.3-2.2.3.1 - On-treatment Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.3.1

#### PROGRAMMING NOTES:

Include all gradable Clinical Chemistry parameters

Table 14.3-2.2.3.2 - On-treatment Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) - Expansion

Replicate of Table 14.3-2.1.3.2

#### PROGRAMMING NOTES:

Include all gradable Clinical Chemistry parameters



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.2.4.1 - Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.4.1

#### PROGRAMMING NOTES:

Include all gradable Clinical Chemistry parameters

Table 14.3-2.2.4.2 - Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.4.2

## PROGRAMMING NOTES:

Include all gradable Clinical Chemistry parameters



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.3.1.1 - Summary of Coagulation Laboratory Data (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.1.1

## PROGRAMMING NOTES:

- Coagulation parameters are PT and aPTT.
- Only Day 1 visit of each cycle

Table 14.3-2.3.1.2 - Summary of Coagulation Laboratory Data (Safety Population) - Expansion

Replicate of Table 14.3-2.1.1.2

#### PROGRAMMING NOTES:

- Coagulation parameters are PT and aPTT.
- Only Day 1 visit of each cycle

Table 14.3-2.3.2.1 - Outside of Normal Range - Shift Table for Coagulation Laboratory Parameters (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.2.1

- Coagulation parameters are PT and aPTT.
- Only Day 1 visit of each cycle.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.3.2.2 - Outside of Normal Range - Shift Table for Coagulation Laboratory Parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.2.2

- Coagulation parameters are PT and aPTT.
- Only Day 1 visit of each cycle.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.4.1.1 - Summary of Thyroid Panel Laboratory Data (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.1.1

## PROGRAMMING NOTES:

- Thyroid Panel parameters are TSH, Free T4 and Free and total T3.
- Only Day 1 visit of each cycle.

Table 14.3-2.4.1.2 - Summary of Thyroid Panel Laboratory Data (Safety Population) - Expansion

## Replicate of Table 14.3-2.1.1.2

#### PROGRAMMING NOTES:

- Thyroid Panel parameters are TSH, Free T4 and Free and total T3.
- Only Day 1 visit of each cycle.

Table 14.3-2.4.2.1 - Outside of Normal Range - Shift Table for Thyroid Panel Laboratory Parameters (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.2.1

- Thyroid Panel parameters are TSH, Free T4 and Free and total T3.
- Only Day 1 visit of each cycle.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.4.2.2 - Outside of Normal Range - Shift Table for Thyroid Panel Laboratory Parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.2.2

- Thyroid Panel parameters are TSH, Free T4 and Free and total T3.
- Only Day 1 visit of each cycle.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Table 14.3-2.5.1 - Summary of Other Laboratory Data (Safety Population) - Dose Escalation

| Visit/<br>Parameter | CPX-POM<br>30 mg/m^2<br>N=X | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| SCR | | | | | | | |
| Pregnancy test? [n (%)] [a] | | | | | | | |
| Negative | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Positive | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| BAS | | | | | | | |
| Pregnancy test? [n (%)][a] | | | | | | | |
| Negative | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Positive | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

[a] Denominator for the percentages was the number of females of child bearing potential.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-2.5.2 - Summary of Other Laboratory Data (Safety Population) - Expansion

Replicate of Table 14.3-2.6.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-3.1.1 - Summary of Vital Signs (Safety Population) - Dose Escalation

Replicate of Table 14.3-2.1.1.1

## PROGRAMMING NOTES:

- Update "laboratory parameter" by "parameter".
- Vital signs include pulse rate, blood pressure, respiratory rate, oxygen saturation and temperature.
- On Days 1 and 5, vital signs are measured at pre-dose and at 6-hour intervals post-dose.

Table 14.3-3.1.2 - Summary of Vital Signs (Safety Population) - Expansion

Replicate of Table 14.3-2.1.1.2

- Update "laboratory parameter" by "parameter".
- Vital signs include pulse rate, blood pressure, respiratory rate, oxygen saturation and temperature.
- On Days 1 and 5, vital signs are measured at pre-dose and at 6-hour intervals post-dose.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-3.2.1 - Summary of Abnormal Vital Signs (Safety Population) - Dose Escalation

| Parameter/<br>Visit/ | CPX-POM 30 mg/m^2 N=X | CPX-POM [D2] mg/m^2 N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM [D6] mg/m^2 N=X | CPX-POM [D7] mg/m^2 N=X |
|---|---|---|---|---|---|---|---|
| Category | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Pulse rate (bpm) [b] | | | | | | | |
| BAS [a] * | XX | XX | XX | XX | XX | XX | XX |
| > 150 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [101-150] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 55 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| C1 TRT D2 * | XX | XX | XX | XX | XX | XX | XX |
| > 150 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [101-150] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 55 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

## <repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>
<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

<sup>\*</sup> Total number of abnormal results at each visit, used as the denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>[</sup>b] Pulse rate: > 150 bpm: Very High values; [101-150] bpm: High values; < 55 bpm: Low values.

<sup>[</sup>c] Systolic Blood Pressure: >= 161 mmHg: Very High values; [131-160] mmHg: High values; < 95 mmHg: Low values.

<sup>[</sup>d] Diastolic Blood Pressure: >= 101 mmHg: Very High values; [86-100] mmHg: High values; < 50 mmHg: Low values.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Table 14.3-3.2.1 - Summary of Abnormal Vital Signs (Safety Population) - Dose Escalation

| Parameter/<br>Visit/<br>Category | | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM<br>[D4] mg/m^2<br>N=X<br>n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|---|
| Systolic Blooc | (mmHg) [c] | | | | | | | |
| BAS [a] * | | XX | XX | XX | XX | XX | XX | XX |
| >= 161 mmF | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [131-160] mmHg | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 95 mmHg | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| C1 TRT D2 * | | XX | XX | XX | XX | XX | XX | XX |
| >= 161 mmF | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [131-160] | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 95 mmHg | | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

## <repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>

<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>\*</sup> Total number of abnormal results at each visit, used as the denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>[</sup>b] Pulse rate: > 150 bpm: Very High values; [101-150] bpm: High values; < 55 bpm: Low values.

<sup>[</sup>c] Systolic Blood Pressure: >= 161 mmHg: Very High values; [131-160] mmHg: High values; < 95 mmHg: Low values.

<sup>[</sup>d] Diastolic Blood Pressure: >= 101 mmHq: Very High values; [86-100] mmHq: High values; < 50 mmHq: Low values.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-3.2.1 - Summary of Abnormal Vital Signs (Safety Population) - Dose Escalation

| Parameter/<br>Visit/<br>Category | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D2] mg/m^2<br>N=X<br>n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Diastolic Blood Pressure (mmHg) [d] | | | | | • | | · · |
| BAS [a] * | XX | XX | XX | XX | XX | XX | XX |
| >= 101 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [86-100] mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 50 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| C1 TRT D2 * | XX | XX | XX | XX | XX | XX | XX |
| >= 101 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [86-100] mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 50 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

## <repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>
<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.

<sup>\*</sup> Total number of abnormal results at each visit, used as the denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>[</sup>b] Pulse rate: > 150 bpm: Very High values; [101-150] bpm: High values; < 55 bpm: Low values.

<sup>[</sup>c] Systolic Blood Pressure: >= 161 mmHg: Very High values; [131-160] mmHg: High values; < 95 mmHg: Low values.

<sup>[</sup>d] Diastolic Blood Pressure: >= 101 mmHg: Very High values; [86-100] mmHg: High values; < 50 mmHg: Low values.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-3.2.2 - Summary of Abnormal Vital Signs (Safety Population) - Expansion

Replicate of Table 14.3-3.2.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-4.1.1 - Summary of ECG Parameters (Safety Population) - Dose Escalation

## Replicate of Table 14.3-2.1.1.1

## PROGRAMMING NOTES:

- Update "laboratory parameter" by "ECG parameter".
- ECG parameters include Heart Rate, PR Interval, RR interval, QRS Duration, QT Interval, QTcF Interval.

Table 14.3-4.1.2 - Summary of ECG Parameters (Safety Population) - Expansion

Replicate of Table 14.3-2.1.1.2

- Update "laboratory parameter" by "ECG parameter".
- ECG parameters include Heart Rate, PR Interval, RR interval, QRS Duration, QT Interval, QTcF Interval.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----

Page X of Y

Table 14.3-4.2.1 - Summary of Abnormal ECG Intervals (Safety Population) - Dose Escalation

| Parameter/<br>Visit/<br>Category | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM<br>[D5] mg/m^2<br>N=X<br>n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| QTcF interval (msec) | | | | | | | |
| BAS [a]* | XX | XX | XX | XX | XX | XX | XX |
| > 450 msec<br>> 480 msec<br>> 500 msec (CS) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) |
| C1 TRT D5 * | XX | XX | XX | XX | XX | XX | XX |
| > 450 msec<br>> 480 msec<br>> 500 msec | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X) XX (XXX.X) XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X)<br>XX (XXX.X) |
| Change from Baseline to C1 TRT D5 * | XX | XX | XX | XX | XX | XX | XX |
| > 30 msec<br>> 60 msec (CS) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) | XX (XXX.X)<br>XX (XXX.X) |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit>
<for last cycle, repeat for Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>\*</sup> Total number of abnormal results at each visit, used as the denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment. CS = Clinically Significant; NCS = Not Clinically Significant.


**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----

Page X of Y

Filename: (Specify file name.rtf)

## Table 14.3-4.2.1 - Summary of Abnormal ECG Intervals (Safety Population) - Dose Escalation

| Parameter/<br>Visit/<br>Category | CPX-POM<br>30 mg/m^2<br>N=X<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| PR interval | | | | | | | |
| Percent Change from Baseline to C1 TRT D5 * | XX | XX | XX | XX | XX | XX | XX |
| ≥ 50% increase from baseline if baseline < 200 ms | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| $\geq$ 25% increase from baseline if baseline $\geq$ 200 ms | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| QRS duration | | | | | | | |
| Percent Change from Baseline to C1 TRT D5 * | XX | XX | XX | XX | XX | XX | XX |
| ≥ 50% increase from baseline if baseline < 110 ms | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| $\geq$ 25% increase from baseline if baseline $\geq$ 110 ms | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

## <for Cycle 2 to last-1 cycle, repeat for Day 1 visit> <for last cycle, repeat for Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.

 $<sup>^{\</sup>star}$  Total number of abnormal results at each visit, used as the denominator for the percentages.

 $<sup>\</sup>hbox{\tt [a] Baseline was the last value/result of assessment prior to or on day of first study treatment.}$ 

CS = Clinically Significant; NCS = Not Clinically Significant.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-4.2.2 - Summary of Abnormal ECG Intervals (Safety Population) - Expansion

Replicate of Table 14.3-4.2.1

### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Table 14.3-4.3.1 - Shift Table for ECG Overall Interpretation (Safety Population) - Dose Escalation

Dose group :  $CPX-POM 30 mg/m^2 (N=X)$ 

| | | Baseline [a] value |
|---|---|---|
| | Value | Abnormal, CS n Abnormal, |
| Visit | at Visit | Normal n (%) (%) NCS n (%) Total |
| C1 TRT D5 (N*=XX) | Normal | XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| | Abnormal, CS | $XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X)$ |
| | Abnormal, NCS | $XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X)$ |
| | Total | XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| C2 TRT D1 (N*=XX) | Normal | XX (XXX.X) XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| | Abnormal, CS | XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| | Abnormal, NCS | $XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X)$ |
| | Total | XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| C2 TRT D5 (N*=XX) | Normal | XX (XXX.X) XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| | Abnormal, CS | $XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X) \qquad XX (XXX.X)$ |
| | Abnormal, NCS | XX (XXX.X) XX (XXX.X) XX (XXX.X) |
| | Total | XX (XXX.X) XX (XXX.X) XX (XXX.X) XX (XXX.X) |

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 5 visit>
<for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit>
<repeat for all doses groups>

Percentage was based on the number of patients present at each visit with non-missing results for the ECG overall interpretation.

\* Denominator of the percentage.

[a] Baseline was the last value of assessment prior to or on day of first study treatment intake.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Repeat for all doses groups, including 'CPX-POM All Doses'.



**Statistical Analysis Plan (TFL shells):** 


Table 14.3-4.3.1 - Shift Table for ECG Overall Interpretation (Safety Population) - Expansion

Replicate of Table 14.3-4.3.1

### PROGRAMMING NOTES:

• Include three columns for 'Cisplatin ineligible', 'Chemotherapy eligible', 'Overall'.



Statistical Analysis Plan (TFL shells):


## **Figures**

Figure 14.2-4.2 - Recurrence-Free Survival (RFS) (Efficacy Population) - Expansion



#### PROGRAMMING NOTES:

- Add legend for group labels accordingly: 'Cisplatin ineligible', 'Chemotherapy eligible'.
- X-axis Label "Recurrence-free survival (months)", Y-axis Label "Survival probability (%)."
- Legend: "Median" and 95% CI.
- Flag censored observations with '+' and add legend.
- If the median time to event has not been reached, present as "Median (95% CI) NR (xx.x, xx.x)" [replacing xx.x with '- ' if there is no upper or lower confidence limit] and add footnote: NR = Median time not reached.



**Statistical Analysis Plan (TFL shells):** 


Figure 14.2-5.2 - Overall Survival (OS) (Efficacy Population) - Expansion

Replicate of Figure 14.2-4.2

### PROGRAMMING NOTES:

• Replace 'Recurrence-Free Survival' by 'Overall Survival' in the figure.



**Statistical Analysis Plan (TFL shells):** 


## Listings

Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.1-1.1.1 - Preface to Inclusion and Exclusion Criteria - Dose Escalation

| Protocol | Inclusion/ | |
|---|---|---|
| Version | Exclusion No. | . Inclusion / Exclusion Text |
| 2 0 | | |
| 3.0 | INCL01 | Patient has histologically- or cytologically- confirmed metastatic or advanced-stage solid malignant tumor that is refractory to standard therapy. Patients should only be included if no therapy exists or if they have received all standard therapies that would be potentially curative or might provide significant benefit. |
| | INCL02 | Patient may have received up to 4 prior lines of cytotoxic chemotherapy or immunotherapy for their metastatic disease (e.g., docetaxel + doxorubicin ± cyclophosphamide), and also may have received additional prior endocrine therapy, as appropriate (e.g., for breast or prostate cancer), or non-myelosuppressive therapy (e.g., bevacizumab, trastuzumab). |
| | <etc></etc> | |
| | EXCL01 | Patient has a history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome) or requires the use of concomitant medications that prolong the QT/QTc interval during study participation. |
| | EXCL02 | Patient has an abnormal cardiac appearance/heart size, as evidenced by chest X-ray or computed tomography (CT) scan. |
| | <etc></etc> | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- List all Inclusion / Exclusion criteria as per eCRF.
- Note: Inclusion / Exclusion text displayed in the listing shell is based on the text in Protocol Version 3.0, but all Inclusion / Exclusion criteria for each of the protocol version (initial to last) should be listed.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.1-1.1.2 - Preface to Inclusion and Exclusion Criteria - Expansion

Replicate of Listing 16.2.1-1.1.1

### PROGRAMMING NOTES:

- List all Inclusion / Exclusion criteria as per eCRF.
- Note: as expansion has been added in PA5, all Inclusion / Exclusion criteria for each of the protocol version from PA5 should be listed.
- Add footnote: Expansion has been added to the protocol from version 5.0.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.1-1.2.1 - List of Failed Inclusion and Exclusion Criteria
(All Patients) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Protocol<br>Version | Failed Inclusion / Exclusion |
|---|---|---|---|
| XXXX | [D3] mg/m^2 | 3.0 | INCL01 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | [D5] mg/m^2 | 3.0 | INCL02 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

## <to be completed with the other patients having at least one protocol deviation>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- List all Inclusion / Exclusion criteria that are failed (i.e. 'N' for inclusion and 'Y' for exclusion)
- Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.1-1.2.2 - List of Failed Inclusion and Exclusion Criteria (All Patients) - Expansion

## Replicate of Listing 16.2.1-1.2.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.1-2.1 - Patient Disposition (Safety Population) - Dose Escalation

| Center/<br>Patient | Country | CPX-POM<br>Dose group | Did the patient complete a full cycle (including Day 22 assessments) and the Follow Up Visit? | Date (day) of<br>Discontinuation/<br>Completion | Reason for<br>Discontinuation,<br>specify | Date<br>(day) of<br>Last Dose | Date (day)<br>of Death | Reason<br>for Death |
|---|---|---|---|---|---|---|---|---|
| XXXX | XXX | 30 mg/m^2 | Yes | DDMMMYYYY (XXX) | | DDMMMYYYY<br>(XXX) | | |
| XXXX | XXX | [D2] mg/m^2 | Yes | DDMMMYYYY (XXX) | | DDMMMYYYY<br>(XXX) | | |
| XXXX | XXX | [D3] mg/m^2 | Yes | DDMMMYYYY (XXX) | | DDMMMYYYY<br>(XXX) | | |
| XXXX | XXX | [D4] mg/m^2 | Yes | DDMMMYYYY (XXX) | | DDMMMYYYY<br>(XXX) | | |
| XXXX | XXX | [D4] mg/m^2 | No | DDMMMYYYY (XXX) | Adverse Event | DDMMMYYYY | | |
| XXXX | XXX | [D4] mg/m^2 | Yes | DDMMMYYYY (XXX) | | (XXX)<br>DDMMMYYYY<br>(XXX) | | |

### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Listing 16.2.1-2.2 - Patient Disposition (Safety Population) - Expansion

| Center/<br>Patient | Country | Group | Completed end of<br>Treatment Visit (Day<br>42 or Day 64)/<br>Reason for Treatment<br>Discontinuation | Date (day) of<br>Treatment Visit<br>Completion /<br>Discontinuation | Date (day) of<br>Last Dose | Date (day) of<br>End of Study | Reason for<br>End of Study |
|---|---|---|---|---|---|---|---|
| XXXX | XXX | Cisplatin ineligible | Yes | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | | |
| XXXX | XXX | Chemotherapy eligible | Yes | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | Lost to Follow up |
| XXXX | XXX | Chemotherapy eligible | Yes | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | | |
| XXXX | XXX | Cisplatin ineligible | Yes | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | | |
| XXXX | XXX | Chemotherapy eligible | No / Adverse Event | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | Withdrawn<br>Consent |
| XXXX | XXX | Cisplatin ineligible | Yes | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | | |
| <0+a> | | | | | | | |

#### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.2.1 - Protocol Deviations (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | - <del></del> | | Leading to Exclusion from Analysis Population(s) | Classification | |
|---|---|---|---|---|---|---|
| XXXX | [D4] mg/m^2 | Compliance | Not treated | xxxxxxx | Safety / Efficacy | • |

## <to be completed with the other patients having at least one protocol deviation>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.2.2 - Protocol Deviations (Safety Population) - Expansion

Replicate of Listing 16.2.2.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.3.1 - Analysis Populations (Safety Population) - Dose Escalation

| Center/<br>Patient | Country | CPX-POM<br>Dose group | Safety Population | Efficacy Population |
|---|---|---|---|---|
| XXXX | XXX | 30 mg/m^2 | Yes | Yes |
| XXXX | XXX | [D2] mg/m^2 | Yes | Yes |
| XXXX | XXX | [D3] mg/m^2 | Yes | No |
| XXXX | XXX | [D4] mg/m^2 | Yes | Yes |
| XXXX | XXX | [D4] mg/m^2 | No | No |
| XXXX | XXX | [D4] mg/m^2 | Yes | Yes |

#### <etc>

The safety population consists of all patients who received at least one dose of CPX-POM.

The efficacy population consists of all patients who have received at least one dose of CPX-POM, had RECIST measurable disease at baseline and had at least one other post-baseline tumor assessment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

• Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.3.2 - Analysis Populations (Safety Population) - Expansion

Replicate of Listing 16.2.3.1

#### PROGRAMMING NOTES:

- Replace definition of efficacy population in footnote by 'The Efficacy population consists of all patients who have received at least one dose of CPX-POM and had tumor tissue at baseline and at the time of RC.'
- Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'/'Chemotherapy eligible'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Listing 16.2.4-1.1 - Demographic and Baseline Characteristics (Safety Population) - Dose Escalation

| Center/<br>Patient | Country | CPX-POM<br>Dose group | Age<br>(year) | Sex | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m^2) | BSA<br>(kgxm) | Female of Child Bearing Potential? | ECOG<br>[a] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXX | 30 mg/m^2 | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D2] mg/m^2 | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | Yes | XXX |
| XXXX | XXX | [D3] mg/m^2 | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | No | XXX |
| XXXX | XXX | [D4] mg/m^2 | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D4] mg/m^2 | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D4] mg/m^2 | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | No | XXX |

#### <etc>

Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Age was calculated from date of birth and date of screening. BMI  $(kg/m^2)$  = Weight (kg) /Height  $(m)^2$ . BSA (kgxm) = 0.007184 x Weight  $(kg)^0$ .425 x (Height  $(cm)^0$ .725 (Dubois formula).

[a] 0 = Fully active. Able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light house work and office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited selfcare. Confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.4-1.2 - Demographic and Baseline Characteristics (Safety Population) - Expansion

Replicate of Listing 16.2.4-1.1

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-2.1 - Pregnancy Test Results (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Visit | Parameter | Assessment Performed? | Assessment<br>Date | Study<br>Day | Result |
|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | SCR | Pregnancy Test | Yes | DDMMMYYYY | XX | Negative |
| | | BAS | Pregnancy Test | Yes | DDMMMYYYY | XX | Positive |

## <repeat for Day 1 of next cycles if relevant> <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Only females are included in this listing.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

• Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.4-2.2 - Pregnancy Test Results (Safety Population) - Expansion

### Replicate of Listing 16.2.4-2.1

### PROGRAMMING NOTES:

• Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'.'



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-3.1 - Cancer History (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Primary Tumor<br>Type | Initial Histological<br>or Cytological<br>Diagnosis<br>Date (Day) | Disease<br>Stage at<br>Screening | Presence of Metastases? | Location |
|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | XXXXX | DDMMMYYYY (XXX) | Grade X | No | |
| XXXX | [D2] mg/m^2 | XXXXX | DDMMMYYYY (XXX) | Grade X | No | |
| XXXX | [D3] mg/m^2<br>[D4] mg/m^2 | XXXXX<br>XXXXX | DDMMMYYYY (XXX) | Grade X<br>Grade X | Yes<br>No | Adrenals/ Bone |
| XXXX | [D4] mg/m^2 | Other, XXXXX | DDMMMYYYY (XXX) | Grade X | Yes | Liver/ Other, XXXXX |
| XXXX | [D4] mg/m^2 | XXXXX | YYYY | Grade X | Yes | Lungs |

### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Listing 16.2.4-4.1 - Prior Cancer Therapies (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Therapy<br>Type | Therapy<br>Name | Line of<br>Therapy | Treatment<br>Setting | Treatment<br>Intent | Start Date (Day)/<br>End Date (Day) | Best<br>Response | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | XXXXX | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX) /<br>DDMMMYYYY (XX) | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | XXXXX | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX) / DDMMMYYYY (XX) | XXXXX | XXXXX |
| XXXX | [D3] mg/m^2 | Radiation,<br>XXXXX | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX) / DDMMMYYYY (XX) | XXXXX | XXXXX |

#### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-5.1 - Medical History and Concomitant Disease (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date (Day) | End Date (Day) | Any medication/non-<br>drug therapies<br>currently being<br>taken for this<br>condition? |
|---|---|---|---|---|
| XXXX | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXXX | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | No |
| XXXX | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXX | MMMYYYY | Ongoing | Yes |

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

MedDRA <version no.>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.4-5.2 - Medical History and Concomitant Disease (Safety Population) - Expansion

Replicate of Listing 16.2.4-5.1

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-6.1 - Cardiac Function (Safety Population) - Dose Escalation

| Center/P<br>atient | CPX-POM<br>Dose group | Visit | Echocardiogra<br>m or MUGA<br>Scan<br>performed? | Method of<br>Assessment | Date of<br>Assessment | Left ventricula r ejection fraction (%) | Overall<br>Interpretatio<br>n | If Clinically<br>Significant,<br>specify |
|---|---|---|---|---|---|---|---|---|
| | | | | Echocardiogra | | | | |
| XXXX | 30 mg/m^2 | C1 TRT D1 | Yes | m | DDMMMYYYY | XX | XXXXX | |
| XXXX | [D2] mg/m^2 | C1 TRT D1 | Yes | MUGA | DDMMMYYYY | XX | Abnormal CS | XXXXX |
| | | | | Echocardiogra | | | | |
| XXXX<br><etc></etc> | [D3] mg/m^2 | C1 TRT D1 | Yes | m | DDMMMYYYY | XX | XXXXX | |

NCS: Not Clinically Significant; CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.4-6.2 - Cardiac Function (Safety Population) - Expansion

## Replicate of Listing 16.2.4-6.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-7.1 - Ophthalmologic Exam (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Visit | Ophthalmology<br>Assessments<br>performed? | Assessment performed by a qualified Ophthalmologist? | Use of<br>Corrective<br>Lenses? | Date of<br>Assessment | Overall<br>Interpretation | If Abnormal CS, specify |
|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 | Yes | Yes | Yes | DDMMMYYYY | XXXXX | |
| XXXX | [D2] mg/m^2 | C1 TRT D1 | Yes | No | No | DDMMMYYYY | Abnormal CS | XXXXX |
| XXXX | [D3] mg/m^2 | C1 TRT D1 | Yes | Yes | No | DDMMMYYYY | XXXXX | |
| <etc></etc> | | | | | | | | |

NCS: Not Clinically Significant; CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Listing 16.2.4-8.1.1 - Prior and Concomitant Medications (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Category | Therapeutic Class<br>Preferred Term<br>Verbatim | Start Date (Day)/<br>End Date (Day) | Dose (unit)/<br>Frequency/<br>Route | Prophylaxis?/<br>Reason |
|---|---|---|---|---|---|
| XXXX | Prior | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXX | DDMMMYYYY (-180)/<br>DDMMMYYYY (XXX) | XXXXXXXX (XXX)/<br>Once/<br>Inhalation | Yes/ XXXXXXXXXXXX |
| | Conc. | XXXXXX/<br>XXXXXXXXXXXX<br>XXXXXXXXXXX | MMMYYYY/<br>Ongoing | Other, XXXX/<br>bid/<br>Cutaneous | No/ XXXXXX |
| XXXX | Prior | XXXXXX/<br>XXXXXXXXXXXX | MMMYYYY/<br>DDMMMYYYY (XXX) | 200 mg/<br>tid/<br>Other, XXXXX | Yes/<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Prior = any medication whose end date is before the date of first dose.

Conc. = concomitant = any medication that started before the date of first dose and stopped on (or is ongoing after) the date of first dose OR any medication whose start date is either the same as (or after) the date of first dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Listing to be sorted by increasing CPX-POM dose.
- Use abbreviations or codes to present data if not enough space (and add appropriate abbreviations / codes in footnotes).



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.4-8.1.2 - Prior and Concomitant Medications (Safety Population) - Expansion

Replicate of Listing 16.2.4-8.1.1

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.4-8.2.2 - Chemotherapy (Safety Population) - Expansion

| Center/<br>Patient | Name of<br>Medication | Start Date (Day)/<br>End Date (Day) | Dose (unit)/<br>Route |
|---|---|---|---|
| XXXX | Gemcitabine<br>Cisplatin | DDMMMYYYY (XXX)/ DDMMMYYYY (XXX)MMMYYYY/ Ongoing | XXXXXXXX (XXX) / XXXXXXXXX (XXX) / XXXXXXXXX |
| XXXX | xxxxxxx | MMMYYYY/<br>DDMMMYYYY (XXX) | XXXXXXXX (XXX) /<br>XXXXXXXX |

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Only patients from Chemotherapy eligible group are included in this listing.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001 --- DELIVERY TYPE --- Extract date: DDMMMYYYY


Listing 16.2.4-9.1 - Surgeries and Procedures (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

System Organ Class/
Center/ Preferred Term/
Patient Verbatim Start Date (Day)

XXXX XXXXXX/ DDMMMYYYY (XXX)

XXXXX/

XXXXXXXXXX

XXXX XXXXX/ --MMMYYYY

XXXXX/

XXXXXXXXXX

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

MedDRA <version no.>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.4-9.2 - Surgeries and Procedures (Safety Population) - Expansion

Replicate of Listing 16.2.4-9.1

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Listing 16.2.5-1.1 - Treatment Administration (Safety Population) - Dose Escalation

| Center/<br>Patient | Visit | CPX-POM<br>Dose<br>group | CPX-POM Dose Amount per Protocol?/ If no, Reason for Adjustment? | Total Infusion Bag Volume of Saline and CPX- POM (ml) | Was Total Volume Infused?/ If no, actual Volume Infused (ml)? | Administration<br>Date (Day)<br>Infusion Start<br>Time- End Time | Arm Used<br>for IV | Infusion<br>Interrupted? |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX | BAS | 30 mg/m^2 | Yes | XXX | Yes | DDMMMYYYY (XX)<br>HH:MM-HH:MM | Right | |
| | C1 TRT<br>D2 | 30 mg/m^2 | Yes | XXX | Yes | DDMMMYYYY (XX)<br>HH:MM-HH:MM | Right | |
| | C1 TRT<br>D3 | 30 mg/m^2 | Yes | XXX | Yes | DDMMMYYYY (XX)<br>HH:MM-HH:MM | Right | |
| | C1 TRT<br>D4 | 30 mg/m^2 | Yes | XXX | Yes | DDMMMYYYY (XX)<br>HH:MM-HH:MM | Right | |
| | C1 TRT<br>D5 | 30 mg/m^2 | No/<br>Adverse event | XXX | No/<br>XXX | DDMMMYYYY (XX)<br>HH:MM-HH:MM | Right | Yes [a] |

## <repeat for Days 1,2,3,4 and 5 of next cycles if relevant>

IV: Intravenous.

[a] See further details regarding infusion interruption in Listing 16.2.5-2.1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.5-1.2 - Treatment Administration (Safety Population) - Expansion

Replicate of Listing 16.2.5-1.1

### PROGRAMMING NOTES:

- Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'/'Chemotherapy eligible'.
- In footnote [a], replace 'Listing 16.2.5-2.1' by 'Listing 16.2.5-2.2'.



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.5-2.1 - Infusion Interruption (Safety Population) - Dose Escalation

| Center/<br>Patient | Visit | CPX-POM<br>Dose group | Reason for Infusion Interrupted? | Administration Date (Day) Time Infusion Interrupted | Infusion<br>Restarted? | Time<br>Infusion<br>Restarted | Reason<br>for Not<br>Restarting? | Infusion Site<br>Reaction? |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | C1 TRT D5 | 30 mg/m^2 | Infusion reaction | DDMMMYYYY (XX)<br>HH:MM | No | | Other, XXXXX | Yes |
| XXXXXXXX | C2 TRT D2 | 30 mg/m^2 | Other, XXXXX | DDMMMYYYY (XX)<br>HH:MM | Yes | нн:мм | | No |
| <cont></cont> | | | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- Listing to be sorted by increasing CPX-POM dose.
- Include only patients with infusion interruption.

Listing 16.2.5-2.2 - Infusion Interruption (All Patients Enrolled) - Expansion

## Replicate of Listing 16.2.5-2.1

### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Extract date: DDMMMYYYY

**Sponsor**: CicloMed **Protocol**: CPX-POM-001

Statistical Analysis Plan (TFL shells):


--- DELIVERY TYPE ----


Listing 16.2.5-3.1 - Drug Exposure (Safety Population) - Dose Escalation

| Center/<br>Patient | CPX-POM Dose<br>group | Date of<br>first dose administration | Visit of<br>last dose<br>administration | Date of<br>last dose<br>administration | Exposure<br>(days) | Exposure (mg) |
|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | DDMMMYYYY | C1 TRT D5 | DDMMMYYYY | XX | XX |
| XXXX | [D2] mg/m^2 | DDMMMYYYY | C2 TRT D5 | DDMMMYYYY | XX | XX |

### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMYYYYY.

The CPX-POM exposure expressed in days is defined as: (last dose taken date - first dose taken date +1) + 16 days.

The CPX-POM exposure expressed in mg is defined as: sum of all (dose per m^2 x Body Surface Area), using Body Surface Area calculated at baseline for Cycle 1 and Cycle 2 dose administrations, and calculated on Day 1 of every other treatment cycle

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

from Cycle 3 dose administration.

• Listing to be sorted by increasing CPX-POM dose.

Listing 16.2.5-3.2 - Drug Exposure (Safety Population) - Expansion

Replicate of Listing 16.2.5-3.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Listing 16.2.6-1.1 - RECIST Target Lesions (Efficacy Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Visit/<br>Target Lesions<br>Identified at<br>Screening Visit? | Date of<br>Scans<br>review | Lesion<br>Number | Organ<br>Site | Specific<br>Location<br>within the<br>Organ Site | Lymph<br>Node<br>Type | Method | Lesion<br>Diameter<br>(mm) | Split or coalesced? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | T02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C2 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | DDMMMYYYY | T02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C2 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C3 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

### <etc>

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.6-2.1 - RECIST Non-Target Lesions (Efficacy Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose<br>group | Visit/<br>Non-Target Lesions<br>Identified at Screening<br>Visit? | Date of Scans review | Lesion<br>Number | Organ<br>Site | Specific<br>Location<br>within the<br>Organ Site | Lymph<br>Node<br>Type | Method |
|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT02 | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2]<br>mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |
| | 3 | C2 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT02 | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT03 | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2]<br>mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |
| | - | C2 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C3 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX |

### <etc>

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


## Listing 16.2.6-3.1 - RECIST response (Efficacy Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Visit | Sum of diameters (mm) | Target Lesion<br>Response | Non-Target Lesion<br>Response | Unequivocal new lesions | Overall<br>Response |
|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 | DDMMMYYYY | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1<br>C2 TRT D1 | DDMMMYYYY<br>DDMMMYYYY | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 C2 TRT D1 C3 TRT D1 | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XXXXX<br>XXXXX | XXXXX<br>XXXXX | XXXXX<br>XXXXX | XXXXX<br>XXXXX |

#### <etc>

CR = Complete response; PR = Partial response; SD = Stable disease; PD = Progressive disease; NE = Not evaluable. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.6-4.1 - Tumor Marker (Efficacy Population) - Dose Escalation

| Center/<br>Patient | CPX-POM<br>Dose group | Visit | Tumor marker assessment performed? | Date of assessment | Type of sample | Tumor marker | If other, specify | Result | Unit |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 | Yes | DDMMMYYYY | XXXXX | XXXXX | | XX.X | XXX |
| | | | | | XXXXX | XXXXX | | XX.X | XXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 | Yes | DDMMMYYYY | XXXXX | XXXXX | | XX.X | XXX |
| | | C2 TRT D1 | Yes | DDMMMYYYY | XXXXX | XXXXX | | XX.X | XXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1<br>C2 TRT D1 | Yes<br>No | DDMMMYYYY | XXXXX | Other | XXXXX | XX.X | XXX |
| | | C3 TRT D1 | Yes | DDMMMYYYY | XXXXX | XXXXX | | XX.X | XXX |

### <etc>

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Listing 16.2.6-5.2 - Evaluable TURBT Results (Efficacy Population) - Expansion

| Center/<br>Patient | Group | TURBT performed within 8 weeks prior to cycle 1 Day 1? | Initial<br>or repeat<br>TURBT | Date of<br>procedure | Tumor tissue sample obtained from a referring institution? | Tumor<br>tissue<br>sample<br>obtained<br>from<br>TURBT? | Highest<br>Viable<br>Tumor<br>content in<br>TURBT (%) | Pathological confirmation of Muscularis Propria Invasion? | Archived<br>tumor<br>tissue from<br>TURBT used? |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cisplatin<br>ineligible | Yes | Initial | DDMMMYYYY | Yes | Yes | XX | Yes | Yes |
| XXXX | Chemotherapy eligible | Yes | Repeat | DDMMMYYYY | Yes | No | | Yes | Yes |
| XXXX | Cisplatin ineligible | No | | | | | | | |

### <etc>

TURBT = Transurethral resection of bladder tumour.

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.6-6.2 - Radical Cystectomy (Efficacy Population) - Expansion

| Center/<br>Patient | Group | Formalin-fixed, paraffin-<br>embedded bladder tumor tissue<br>obtained at time of RC | Date of procedure | Tumor tissue sample obtained from cystectomy used? | Highest Viable Tumor content from cystectomy (%) |
|---|---|---|---|---|---|
| XXXX | Cisplatin<br>ineligible | Yes | DDMMMYYYY | Yes | XX |
| XXXX | Chemotherapy eligible | Yes | DDMMMYYYY | No | |
| XXXX | Cisplatin ineligible | Yes | | | |

#### <etc>

RC = Radical cystectomy.

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


# Listing 16.2.6-7.2 - Determination of Recurrence and Survival (Efficacy Population) - Expansion

| Center/<br>Patient | Group | Attend any follow-up visits (includes phone calls)? | If no,<br>reason | Date of<br>Death | Cause of<br>Death | Physician<br>Decision,<br>specify | Other,<br>specify | Date of<br>study<br>completion | Date of last<br>contact with<br>patient |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cisplatin<br>ineligible | No | Death | DDMMMYYYY | XXXXXX | | | DDMMMYYYY | DDMMMYYYY |
| XXXX | Chemotherapy eligible | Yes | | | | | | DDMMMYYYY | DDMMMYYYY |
| XXXX | Cisplatin ineligible | No | Physician<br>Decision | | | XXXXXX | | DDMMMYYYY | DDMMMYYYY |
| XXXX | Cisplatin ineligible | No | | | | | | DDMMMYYYY | DDMMMYYYY |

#### <etc>

Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.6-8.2 - Recurrence-Free Survival and Overall Survival (Efficacy Population) - Expansion

| Center/<br>Patient | Group | Date of<br>first CPX-<br>POM<br>Infusion<br>(Day) | Date of<br>Recurrence<br>(Day) | Date of<br>Death<br>(Day) | Start Date of<br>First Further<br>Anti-cancer<br>Therapy (Day) | Date of<br>Last<br>Contact<br>(Day) | RFS<br>(month) | Censoring<br>/ Event<br>for RFS | OS<br>(month) | Censoring/<br>Event for<br>OS |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cisplatin<br>ineligible | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | | DDMMMYYYY<br>(XX) | xx.x | Event | XX.X | Event |
| XXXX | Chemotherapy eligible | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | XX.X | Censoring | XX.X | Event |
| XXXX | Cisplatin<br>ineligible | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | | DDMMMYYYY<br>(XX) | XX.X | Event | XX.X | Event |
| XXXX | Cisplatin ineligible | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | | DDMMMYYYY<br>(XX) | XX.X | Censoring | XX.X | Censoring |

#### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

RFS = Recurrence Free Survival, OS = Overall Survival.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.7-1.1 - Dose-Limiting Toxicity (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date (Day)/<br>End Date (Day) | Action Taken/<br>Medication or<br>Therapies Taken? | Outcome/<br>Grade/<br>Relationship | SAE? |
|---|---|---|---|---|---|
| XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (XXX)/<br>DDMMMYYYY (XXX) | None/<br>No | XXXXXXX/<br>Grade 1/<br>Not related | No |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY (XXX)/<br>Ongoing | Dose Adjusted/<br>Yes | Resolved/<br>Grade 3/<br>Definitely related | Yes |
| XXXX | XXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXX | DDMMMYYYY (XXX)/<br>MMMYYYY | | XXXXXXX/<br>XXXXXX/<br>XXXXXXX | No |

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

MedDRA version <version #>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where DLT= Yes.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.7-2.1 - Adverse Events (Safety Population) - Dose Escalation

#### Replicate of Listing 16.2.7-1.1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs.

Listing 16.2.7-2.2 - Adverse Events (Safety Population) - Expansion

Replicate of Listing 16.2.7-2.1

#### PROGRAMMING NOTES:

• Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'/'Chemotherapy eligible'.

Listing 16.2.7-3.1 - Serious Adverse Events (Safety Population) - Dose Escalation

Replicate of Listing 16.2.7-1.1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where SAE = Yes.
- Remove column 'SAE'.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.7-3.2 - Serious Adverse Events (Safety Population) - Expansion

## Replicate of Listing 16.2.7-3.1

#### PROGRAMMING NOTES:

• Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'.'

Listing 16.2.7-4.1 - Adverse Events Leading to Discontinuation (Safety Population) - Dose Escalation

### Replicate of Listing 16.2.7-1.1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where action taken = Drug Withdrawn.

Listing 16.2.7-4.2 - Adverse Events Leading to Discontinuation (Safety Population) - Expansion

## Replicate of Listing 16.2.7-4.1

## PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.7-5.1 - Adverse Events Leading to Death (Safety Population) - Dose Escalation

### Replicate of Listing 16.2.7-1.1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where outcome = Fatal

Listing 16.2.7-5.2 - Adverse Events Leading to Death (Safety Population) - Expansion

Replicate of Listing 16.2.7-5.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Filename: (Specify file name.rtf)

Listing 16.2.8-1.1 - Patients Laboratory Profile: Hematology (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Visit | Assessment_<br>Date Tim | Study<br>e Day | Parameter<br>(Unit) | Normal<br>Range | Result | CTCAE<br>grade | Change<br>from<br>Baseline | CS? |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | BAS | DDMMMYYYY HH: | MM XXX | XXXXXXXX (XXXX) | XXXXXX | XX | Grade 1 | | |
| | C1 TRT D1 | DDMMMYYYY HH: | XXX MM | XXXXXXXX (XXXX) | XXXXXX | XX L/H | Grade 2 | XXXX | |
| | C1 TRT D4 | DDMMMYYYY HH: | XXX MM | XXXXXXXX (XXXX) | XXXXXX | XX L/H | Grade 2 | XXXX | |
| | C1 TRT D10 | DDMMMYYYY HH: | XXX MM | XXXXXXXX (XXXX) | XXXXXX | XX L/H | Grade 3 | XXXX | CS |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit and Day 4 visit if relevant> <for the last cycle, repeat also for Day 22 visit and Day 28 visit>

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Baseline was the last non-missing assessment prior or on the first dose date.

SI units and results presented. L/H = low/high value based upon normal ranges.

 ${\tt R = repeat/unscheduled \ assessments. \ CS = Clinically \ Significant; \ NCS = Not \ Clinically \ Significant; \ ND = Not \ Done.}$ 

Laboratory ranges are based on NCI-CTCAE version 4.03.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• Repeat for the other CPX-POM doses by increasing order.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.8-1.2 - Patients Laboratory Profile: Hematology (Safety Population) - Expansion

## Replicate of Listing 16.2.8-1.1

#### PROGRAMMING NOTES:

• Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'.'

Listing 16.2.8-2.1 - Patients Laboratory Profile: Clinical Chemistry (Safety Population) - Dose Escalation

#### Replicate of Listing 16.2.8-1.1

#### PROGRAMMING NOTES:

• Listing to be sorted by increasing order.

Listing 16.2.8-2.2 - Patients Laboratory Profile: Clinical Chemistry (Safety Population) - Expansion

Replicate of Listing 16.2.8-2.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.8-3.1 - Patients Laboratory Profile: Coagulation (Safety Population) - Dose Escalation

## Replicate of Listing 16.2.8-1.1

#### PROGRAMMING NOTES:

- Listing to be sorted by increasing order.
- Only Day 1 of each cycle.

Listing 16.2.8-3.2 - Patients Laboratory Profile: Coagulation (Safety Population) - Expansion

#### Replicate of Listing 16.2.8-3.1

#### PROGRAMMING NOTES:

• Change label from 'CPX-POM Dose group' to 'Group' and populate with 'Cisplatin ineligible'.'

Listing 16.2.8-4.1 - Patients Laboratory Profile: Thyroid Panel (Safety Population) - Dose Escalation

### Replicate of Listing 16.2.8-1.1

#### PROGRAMMING NOTES:

- Listing to be sorted by increasing order.
- Only Day 1 of each cycle.
- Remove CTCAE column and footnote.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.8-4.2 - Patients Laboratory Profile: Thyroid Panel (Safety Population) - Expansion

Replicate of Listing 16.2.8-4.1

#### PROGRAMMING NOTES:



Statistical Analysis Plan (TFL shells):


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.8-5.1 - Patients Laboratory Profile: Urinalysis (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/ | | Assessm | ent | Study Pa | Parameter | Parameter | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Visit | Date | Time | Day | (Unit) | | Range | Result | CS? |
| XXXX | BAS | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | |
| | C1 TRT D1 | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | |
| | C1 TRT D4 | DDMMMYYYY | HH:MM | XXX | XXXXXXX | (XXXX) | XXXXXX | XX | |
| | C1 TRT D10 | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | CS |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit and Day 4 visit if relevant>
<for the last cycle, repeat also for Day 22 visit and Day 28 visit>

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Baseline was the last non-missing assessment prior or on the first dose date.

R = repeat/unscheduled assessments. CS = Clinically Significant; NCS = Not Clinically Significant; ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

Repeat for the other CPX-POM doses by increasing order.

Listing 16.2.8-5.2 - Patients Laboratory Profile: Urinalysis (Safety Population) - Expansion

## Replicate of Listing 16.2.8-5.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.9-1.1 - Vital Signs (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Visit | Assess<br>Date | sment<br>Time | Study<br>Day | Timepoint | Parameter (unit) | Result | Change from Baseline |
|---|---|---|---|---|---|---|---|---|
| XXXX | BAS | DDMMMYYY | Y HH:MM | XXX | | Pulse Rate (bpm) | XXX L | |
| | | | | | | Respiratory Rate (bpm) | XXX | |
| | | | | | | Systolic BP (mmHg) | XXX | |
| | | | | | | Diastolic BP (mmHg) | XXX | |
| | | | | | | Oxygen Saturation (%) | XXX | |
| | | | | | | Body Weight (kg) | XXX.X | |
| | | | | | | Temperature (C) | XX.X | |
| | | | | | 6 hours | | | |
| | C1 TRT D1 | DDMMMYYY | Y HH:MM | XXX | Post Dose | Pulse Rate (bpm) | XXX H | XX |
| | | | | | | Respiratory Rate (bpm) | XXX | XX |
| | | | | | | Systolic BP (mmHg) | XXX VH | XX |
| | | | | | | Diastolic BP (mmHg) | XXX | XX |
| | | | | | | Oxygen Saturation (mmHg) | XXX | XX |
| | | | | | | Body Weight (kg) | XXX.X | X.X |
| | | | | | | Temperature (C) | XX.X | X.X |

<repeat for Day 3, Day 4, Day 5, Day 6 and Day 10 visits of Cycle 1>
<for Cycle 2 to last-1 cycle, repeat from Day 1 to Day 6 visits if relevant>
<for the last cycle, repeat also for Day 22 visit and Day 28 follow-up visit>

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY. Baseline was the last non-missing assessment prior or on the first dose.

L = Low; H = High; VH = Very High; BP = Blood Pressure; bpm = beats per minute; ND = Not Done.

Pulse Rate: L: <55 bpm; H: 101-150 bpm; VH: >150 bpm.

Systolic BP: L: <95 mmHg; H: 131-160 mmHg; VH: >=161 mmHg.

Diastolic BP: L: <50 mmHg; H: 86-100 mmHg; VH: >=101 mmHg.

R = repeated/ unscheduled assessment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



**Statistical Analysis Plan (TFL shells):** 


#### PROGRAMMING NOTES:

- Include all parameters: blood pressure, respiratory rate, pulse, oxygen saturation, temperature, BSA, BMI and height.
- Repeat for all doses groups

Listing 16.2.9-1.2 - Vital Signs (Safety Population) - Expansion

Replicate of Listing 16.2.9-1.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.9-2.1 - ECG Results (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | 77: _: _ | Assessment Date (Day) | Devemates (unit) | De cult | Channe from bassline |
|---|---|---|---|---|---|
| racient | Visit | (Day) | Parameter (unit) | Result | Change from baseline |
| XXXX | BAS | DDMMMYYYY (XXX) | Heart Rate (bpm) | XXX | XX |
| | | , | PR interval (msec) | XXX | XX |
| | | | RR interval (msec) | XXX | XX |
| | | | QRS duration (msec) | XXX | XX |
| | | | QT interval (msec) | XXX | XX |
| | | | QTcF interval (msec) | XXX | XX |
| | | | Overall Interpretation | Normal | |
| | C1 TRT D5 | DDMMMYYYY (XXX) | Heart Rate (bpm) | XXX ++ | XX * |
| | | | PR interval (msec) | XXX | XX |
| | | | RR interval (msec) | XXX | XX |
| | | | QRS duration (msec) | XXX | XX |
| | | | QT interval (msec) | XXX | XX |
| | | | QTcF interval (msec) | XXX + | XX |
| | | | Overall Interpretation | Abnormal, CS | |

# <for Cycle 2 to last-1 cycle, repeat for Day 1 visit if relevant> <for the last cycle, repeat also for Day 28 follow-up visit>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY. Baseline was the last non-missing assessment prior or on the first dose date.

QTcF: +: >450 msec; ++: > 480 msec; +++: >500 msec; \*: > 30 msec above baseline; \*\*: > 60 msec above baseline.

R = repeated/ unscheduled assessment. CS = Clinically significant; NCS = Not Clinically Significant.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• Repeat for all dose groups.



**Statistical Analysis Plan (TFL shells):** 


Listing 16.2.9-2.2 - ECG Results (Safety Population) - Expansion

Replicate of Listing 16.2.9-2.1

#### PROGRAMMING NOTES:



**Statistical Analysis Plan (TFL shells):** 


Protocol: CPX-POM-001
Extract date: DDMMMYYYY

--- DELIVERY TYPE ----


Listing 16.2.9-3.1 - Digital Holter Monitoring (Safety Population) - Dose Escalation

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Visit | Assessment Start<br>Date Time | Assessment End<br>Date Time | Study<br>Day | Any Alert<br>Flags? | Timepoint | Alert Flag<br>Type | Specify |
|---|---|---|---|---|---|---|---|---|
| XXXX | BAS | DDMMMYYYY HH:MM | DDMMMYYYY HH:MM | xx | Yes | Pre-dose | <pre>&gt; 60 ms increase from baseline Other (specify)</pre> | xxxxx |

•••

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY. Baseline was the last non-missing assessment prior or on the first dose date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Repeat for all dose groups.

# **DocuSign**

**Certificate Of Completion** 

Envelope Id: 58ECCD3CFEAF44899B59B738DF5CCA50

Subject: Please DocuSign: CPX-POM-001 Shells v2.0

Source Envelope:

Document Pages: 125 Signatures: 3 Initials: 0

Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Envelope Originator:

Status: Completed

IP Address: 89.80.168.70

Sent: 03-Nov-2021 | 16:55 Viewed: 03-Nov-2021 | 18:49

Signed: 03-Nov-2021 | 18:50

**Record Tracking** 

Status: Original

03-Nov-2021 | 16:53

Holder:

Location: DocuSign

**Signer Events** 

Signature

**Timestamp** 

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

C379E80D-7E44-4D7C-93C1-912BBD696B8A

Using IP Address: 136.32.172.207

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 03-Nov-2021 | 18:49

ID: ef3f196a-5b0d-4032-9c36-eafdc0970a84

Sent: 03-Nov-2021 | 16:55 Viewed: 03-Nov-2021 | 16:55

Signed: 03-Nov-2021 | 16:56

**Biostatistics** 

Cmed (Clinical Research Services) Limited Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

47FCB0F5-C810-4908-9B4A-6F3E0911DFD3

Using IP Address: 89.80.168.70

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 03-Nov-2021 | 16:55

ID: 3c27fc3d-6459-4085-ad57-54a7ba7926d5

| Signer Events | Signature | Timestamp |
|---|---|---|
| | | Sent: 03-Nov-2021 16:55 |
| | | Viewed: 03-Nov-2021 17:44 |
| Medical Advisor | | Signed: 03-Nov-2021 17:47 |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style<br>Signature ID:<br>24D4E3E8-B54A-42C2-8905-70B3A43C3698<br>Using IP Address: 45.27.88.12 | |
| | With Signing Authentication via DocuSign password | ı |
| | With Signing Reasons (on each tab): | |
| | I approve this document | |
| Electronic Record and Signature Disclosure: | | |

Accepted: 03-Nov-2021 | 17:44 ID: 4c3e7195-80ba-482e-aa94-7741cfe27666

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 03-Nov-2021 16:55<br>03-Nov-2021 17:44<br>03-Nov-2021 17:47<br>03-Nov-2021 18:50 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Discl | Electronic Record and Signature Disclosure | |

## ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Cmed (Clinical Research Services) Limited (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

## All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact Cmed (Clinical Research Services) Limited:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: dataprivacy@cmedresearch.com

# To advise Cmed (Clinical Research Services) Limited of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at dataprivacy@cmedresearch.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from Cmed (Clinical Research Services) Limited

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with Cmed (Clinical Research Services) Limited

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify Cmed (Clinical Research Services) Limited as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Cmed (Clinical Research Services) Limited during the course of your relationship with Cmed (Clinical Research Services) Limited.